CLINICAL TRIAL: NCT04548388
Title: EFFECT of WHOLE BODY VIBRATION on FUNCTIONAL CAPACITY and RESPIRATORY FUNCTIONS IN STROKE INDIVIDUALS: A RANDOMIZED CONTROLLED STUDY
Brief Title: EFFECT of WHOLE BODY VIBRATION on FUNCTIONAL CAPACITY and RESPIRATORY FUNCTIONS IN STROKE INDIVIDUALS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Mehmet Duray, Principal Investigator, Suleyman Demirel University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 60116787-020/45178
Record Dates: First submitted 2020-09-08; First posted 2020-09-14 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Stroke; Respiratory Function Impaired
Keywords: Stroke; Bobath approach; whole body vibration; functional capacity; respiratory function
MeSH Terms: conditions — Stroke; Respiratory Insufficiency; Respiratory Aspiration | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bobath approach (Experimental): Bobath approach
  Interventions: Other: rehabilitation
- whole body vibration (Experimental): whole body vibration
  Interventions: Other: rehabilitation

INTERVENTIONS:
Other: rehabilitation — A specialist physiotherapist in neurological rehabilitation provided the Bobath approach individually to each patients in both groups. Bobath approach included 3 days a week over a total of 12 sessions for four weeks. The Bobath approach consisted of about individual one hour session.
  In addition to the Bobath approach, the subjects in the study group received WBV for 20 minutes a day, 2 days a week. The frequency of the device was increased by 5 Hz every week, starting the treatment with 30 Hz. Whole body vibration application was performed on a platform (Power Plate Pro5®) that provides vertical vibration. Two different practice positions were chosen as standing and semi-squatting. In order to prevent muscle fatigue, the set consisting of 1 minute of application - 1 minute of rest in each position was applied for a total of 10 minutes with 5 repetitions

SUMMARY:
While there is only one study examining the effect of WBV on oxygen consumption and cardiovascular responses in individuals with stroke, no study has been found on the effect of WBV on respiratory capacity and flow volumes and changes in functional capacity due to effort. In this study, it was aimed to investigate whether the WBV treatment protocol determined has an effect on functional capacity and respiratory functions in individuals with stroke.

ELIGIBILITY:
Inclusion Criteria:

* having first hemiplegic stroke history at least for 3 months, being clinically stable could stand for at least 1 minute, could walk independently with or without a walking aids.

Exclusion Criteria:

* having any neurological, psychiatric, orthopedic and unstable cardiovascular and pulmonary conditions other than stroke.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2018-11-17 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Six-minute walking test | 12 months
  functional capacity
microQuark® brand PC-based USB spirometer | 12 months
  respiratory capacity

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Duray, Principal Investigator — Suleyman Demirel University
Locations (1):
- Mehmet Duray, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No